CLINICAL TRIAL: NCT01872390
Title: Start TB Patients on ART and Retain on Treatment: Combination Intervention Package to Enhance Antiretroviral Therapy Uptake and Retention During TB Treatment in Lesotho
Brief Title: Start TB Patients on ART and Retain on Treatment (START Study)
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAK7103; AID-OAA-A-12-00022 (Other: Columbia University)
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Tuberculosis; HIV
Keywords: Lesotho; TB; tuberculosis; HIV; antiretroviral therapy; ART; adherence; combination intervention package; retention
MeSH Terms: conditions — Tuberculosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIP Participants (Experimental): Participants will receive the usual procedures (standard of care) for management of HIV-infected TB patients, and in addition the Combination Intervention Package (CIP) with the programmatic, structural, and psychosocial components.
  Interventions: Other: Combination Intervention Package
- SOC Participants (Other): Participants will receive the usual procedures (standard of care) for management of HIV-infected TB patients. TB and HIV services are fully integrated in a one-stop model, while at hospitals, ART is provided in the TB clinic for TB/HIV coinfected patients.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Combination Intervention Package — CIP will contain programmatic, structural and psychosocial components including: 1) nurse training and mentorship in TB/HIV cotreatment using a clinical algorithm; 2) reimbursement of transportation costs to monthly clinic visits for patients and treatment supporters; 3) health education using a TB and HIV treatment literacy curriculum for patients and treatment supporters; and 4) real-time adherence support using short message service (SMS) text messaging and trained village health workers (VHW). These components were selected for their promise, practicality, and feasibility of implementation and scale-up in HIV programs in diverse settings - in addition to SOC.
  Other Names: CIP
  Arms: CIP Participants
Other: Standard of Care — Usual procedures for management of HIV-infected TB patients will be followed: Three I's training, ART provision to TB patients in integrated clinics, and treatment supporter for TB treatment.
  Other Names: SOC
  Arms: SOC Participants

SUMMARY:
The purpose of the START Study is to identify an effective, cost-effective, acceptable intervention that addresses programmatic, structural and psychosocial barriers to ART initiation and retention during TB treatment, with the ultimate goal of improving health outcomes among HIV-infected TB patients in Lesotho. The study is a two-arm cluster randomized trial, randomized at the TB/HIV clinic level, which includes twelve TB/HIV clinics in Berea district. Clinics are randomized to deliver the combination intervention package (CIP) or standard of care (SOC), with stratification by facility type. The experimental intervention will be delivered to all HIV-infected TB patients in TB/HIV clinics randomly assigned to CIP. In TB/HIV clinics assigned to SOC, usual care procedures for ART initiation and retention will be delivered.

Study hypotheses focus on the effectiveness of the CIP on HIV- and TB-related outcomes.

Compared to HIV-infected TB patients attending SOC clinics, HIV-infected TB patients at CIP clinics will have superior HIV- and TB-related outcomes, including:

* Greater ART initiation during TB treatment
* Shorter time to ART initiation
* Greater retention in ART care
* Higher adherence to ART
* Greater change in CD4+ count
* Greater TB treatment success (completion and cure)
* Greater sputum smear conversion
* Higher adherence to TB treatment

Additionally, CIP delivery will have an incremental cost-effectiveness ratio more favorable than alternative resource uses.

DETAILED DESCRIPTION:
Among people living with HIV (PLWH), tuberculosis (TB) is the most common opportunistic illness and a leading cause of death, accounting for nearly a quarter of HIV-related deaths worldwide. Initiating antiretroviral therapy (ART) early during TB treatment significantly increases survival, and World Health Organization (WHO) guidelines recommend ART initiation for all PLWH as soon as possible after TB treatment initiation, regardless of CD4+ count. Yet in the African Region, only 42% of TB patients known to be living with HIV were on ART in 2010, and retention in ART programs has been limited. In Lesotho, only 27% of HIVinfected TB patients received ART in 2010. There is an urgent need to identify programmatic interventions that increase the proportion of HIV-infected TB patients on ART, shorten the duration between TB diagnosis and ART initiation, and improve adherence to medications and retention in care amongst HIV-infected TB patients in Lesotho.

Lesotho, a small, landlocked country completely surrounded by South Africa, is among the world's poorest nations with one of the world's most severe epidemics of HIV and tuberculosis (TB). There is strong evidence that TB patients who are also infected with HIV have better survival rates if they begin antiretroviral therapy (ART) soon after starting TB treatment; however, there are many patients who do not initiate ART within the recommended timeframe, and who do not remain in care.

ELIGIBILITY:
Measurement Cohort Participant Inclusion Criteria:

1. HIV-infected
2. On TB treatment
3. Initiating ART within 2 months of TB treatment initiation
4. Aged 18 or older
5. English- or Sesotho-speaking
6. Capable of informed consent

Measurement Cohort Participant Exclusion Criteria:

1. Children under age of 18
2. Patients diagnosed with Multi Drug Resistant-TB (MDR-TB)

Key Informats: Three groups of key informats (KI) will be recruited.

* Key Informants ART Early-Initiators Inclusion Criteria:

  1. A measurement cohort participant
  2. Initiaing ART within the first 8 weeks of TB treatment
* Key Informants ART Non/Late-Initiators Inclusion Criteria:

  1. A measurement cohort participant
  2. did not initiate ART during TB treatment or initiating ART >= 2 months after TB treatment initiation
* Key Informants Healthcare Workers Inclusion Criteria:

  1. Nurse or VHW working in a CIP clinic or VHW working in the community and affiliated with CIP clinic
  2. Aged 18 or older
  3. English- or Sesotho-speaking
  4. Capable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Percentage of TB/HIV patients newly registered during period of observation who initiate ART during TB treatment | Up to 9 months
  To examine ART initiation based on review of clinic registers.
Percentage of participants who attended 6 month clinic visit (within 1 month window) and reported ART use | Up to 6 months after TB treatment initiation
  To examine ART retention. Deaths and transfers will be considered not retained.
Participants with cure + treatment completion at end of TB treatment | Up to 9 months
  To examine TB treatment success as defined by WHO, based on review of TB register and treatment cards.

SECONDARY OUTCOMES:
Days from TB treatment initiation to date of ART initiation | Up to 9 months
  To examine Time to ART initiation
Percentage of total prescribed doses ingested for ART | Up to 9 months
  To examine ART adherence, averaged across medicines for each month of treatment, from the unannounced pill counts.
Change in CD4+ count | Up to 6 months after initial CD4 count
  To examine change in CD4 count over 6 months (from initiation of TB treatment to 6 months later). Routine clinical CD4 test results will be used by study staff and no additional blood draw will be required.
Percentage of smear positive pulmonary TB cases that converted to smear negative after eight weeks of treatment | Up to 8 weeks from initiation of TB treatment
  To examine sputum smear conversion
Percentage of total prescribed doses ingested for TB treatment | Up to 9 months
  To examine TB treatment adherence, from unannounced pill counts.
Ratio of the incremental costs of the CIP to incremental effectiveness | Up to 2 years
  To examine incremental cost-effectiveness of CIP (per ART initiation, retention, and TB treatment completion)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea A Howard, MD, Principal Investigator — Columbia University
Locations (12):
- Lesotho (12):
  - Koali Health Center, Koali
  - Maluti Hospital, Mafeteng
  - St. Magdalena Health Center, Mafeteng
  - Khubetsoana Health Center, Maseru
  - Pilot Health Center, Maseru
  - Berea Hospital, Teyateyaneng
  - Good Shepherd Health Center, Teyateyaneng
  - Holy Family Health Center, Teyateyaneng
  - Kolojane Health Center, Teyateyaneng
  - Sebedia Health Center, Teyateyaneng
  - St. David Health Center, Teyateyaneng
  - St. Theresa Health Center, Teyateyaneng

IPD SHARING:
Plan to Share IPD: No